CLINICAL TRIAL: NCT03309384
Title: Intraoperative Monitoring (Parathormone Values and Continuous Neuromonitoring) to Predict Postoperative Complications After Total Thyroidectomy
Brief Title: Intraoperative Monitoring to Predict Postoperative Complications After Thyroidectomy
Acronym: PARACAL
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Laurent BRUNAUD, Professor of Surgery, MD, PhD, Central Hospital, Nancy, France
Other Study IDs: PARACAL; R2016-25 (Registry Identifier: CNIL)
Record Dates: First submitted 2017-09-06; First posted 2017-10-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Endocrine Procedural Complications; Thyroid; Parathyroid; Deficiency; Laryngeal Injury
MeSH Terms: conditions — Thyroid Diseases; Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to evaluate the role of intraoperative continous and intermittent neuromonitoring and intraoperative parathormone (PTH) to predict postoperative nerve morbidity and hypocalcemia.

DETAILED DESCRIPTION:
Intraoperative PTH values and intraoperative continuous neuromonitoring will be collected prospectively in consecutive patients who undergo total thyroidectomy.

Postoperative parathyroid morbidity and recurrent laryngeal nerve morbidity will be evaluated within 1 week after total thyroidectomy and at 1 year postoperatively.

Other postoperative morbidity will be evaluated at 1 year postoperatively using validated classification.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for total thyroidectomy in university of Nancy (University Hospital)

Exclusion Criteria:

* refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients scheduled for total thyroidectomy in university of Nancy (University Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-03-20; Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
intraoperative parathormone values | intraoperative
  parathormone in pg/mL

SECONDARY OUTCOMES:
postoperative hypocalcemia | within 1 week after thyroidectomy
  calcium in mg/L
postoperative hypoparathyroidism | within 1 week after thyroidectomy
  parathormone in pg/mL
permanent postoperative hypocalcemia | at one year after thyroidectomy
  calcium in mg/L
permanent postoperative hypoparathyroidism | at one year after thyroidectomy
  parathormone in pg/mL
laryngeal nerve palsy | during thyroidectomy
  continuous intraoperative neuromonitoring (> 50% baseline values yes/no)
laryngeal nerve palsy | within 1 week after thyroidectomy
  laryngoscopy (normal / palsy)
laryngeal nerve palsy | at one year after thyroidectomy
  laryngoscopy (normal / palsy)
Postoperative complications other than outcomes from 1 to 8 | at one year after thyroidectomy
  Postoperative morbidity classification (using a Clavien-Dindo classification) postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Brunaud, Principal Investigator — CHU NANCY
Locations (1):
- CHU Nancy, Vandœuvre-lès-Nancy, France